CLINICAL TRIAL: NCT02116114
Title: Effects of Aquatic Physical Training Program on Cardiorespiratory Variables in Patients With COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Marlene Aparecida Moreno, pos doctorate, Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13/11
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2011-04

CONDITIONS: Adverse Effects in the Aquatic Exercises
Keywords: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aquatic exercises (Experimental): * 3 times a week
  * heating
  * aerobic training
  * slowdown
  Interventions: Other: Aerobic training
- control group (No Intervention): The control group participated in the study only to usual care , conventional medical treatment orientation about the disease , methods of energy conservation and evaluation.

INTERVENTIONS:
Other: Aerobic training — The program of aquatic exercise training was developed involving the following steps : heating : dynamic stretching exercises aerobic exercises , lasting 10 minutes was performed, aquatic fitness : aerobic training and slowdown. The intensity was prescribed based on the Borg scale score 4-6. Aerobic training was performed at intervals. The duration of aerobic fitness was started with eight 20-minute sessions , progressing to eight sessions of 30 minutes and finished with eight 40-minute sessions. Downturn : global stretching exercises , lasting 10 minutes were performed. During all sessions , the patients were instructed to breath with pursed - lip .
  Arms: Aquatic exercises

SUMMARY:
We have as hypothesis that the aquatic aerobic physical training program can help promote beneficial adaptations on the cardiovascular, respiratory and systemic inflammation variables, functional capacity and quality of life in patients with chronic obstructive pulmonary disease (pulmonary emphysema).

DETAILED DESCRIPTION:
First paragraph

* aquatic aerobic physical training program
* beneficial adaptations

Next paragraph

* cardiovascular
* respiratory
* systemic inflammation
* functional capacity
* quality of life

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD ( GOLD I / II / III / IV rating )
* Clinically stable
* Low level of physical activity , according to the IPAQ ( International Physical Activity Questionnaire )
* Absence of exacerbation in the last three months
* Do not participate in a regular exercise program in the past six months

Exclusion Criteria:

* Diabetes Mellitus
* Endocrine Disorders
* Chronic renal failure
* Liver Diseases
* Other lung diseases or inflammatory diseases associated
* Cardiac
* Use of drugs that prevented physical performance
* Musculoskeletal and neuromuscular changes that make it impossible to run experimental protocols
* Dermatological disorders ( cutaneous fistulas , infected wounds , ringworm skin , varicose ulcers )
* Hypersensitivity to the product used for the treatment of pool water
* Rabies

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in cardiac autonomic modulation by heart rate variability at week 8 | Baseline, Week 8

SECONDARY OUTCOMES:
Change from baseline in quality of life by the Saint George Respiratory Questionnaire at week 8 | Baseline, Week 8

OTHER OUTCOMES:
Change from baseline in systemic inflammation by C-reactive protein at week 8 | Baseline, Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Bruna G Silva, Master, Principal Investigator — Universidade Metodista de Piracicaba